CLINICAL TRIAL: NCT06256458
Title: Multicenter Prospective Registry to Evaluate Use and Outcomes of NanoBone® Bone Graft Substitute in Acute Trauma Patients
Brief Title: Prospective Registry to Evaluate Outcomes of NanoBone® Bone Graft in Acute Trauma
Acronym: ARTIST
Status: Recruiting | Type: Observational
Sponsor: Artoss Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ART001
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: NanoBone® Bone Graft — The surgical technique used by the surgeon and the choice of the specific NanoBone product is or was determined solely by the surgeon and is independent of this observational study.

SUMMARY:
This multicenter prospective patient registry was developed with the aim of documenting how orthopedic surgeons are utilizing the NanoBone products in acute trauma cases along with relevant patient outcomes. These outcomes include radiographic measures such as fracture healing, instrumentation integrity, and clinical outcomes (symptom and function improvement) based on investigator and patient-based outcome assessments.

DETAILED DESCRIPTION:
This multicenter prospective patient registry was developed with the aim of documenting how orthopedic surgeons are utilizing the NanoBone products in acute trauma cases along with relevant patient outcomes. These outcomes include radiographic measures such as fracture healing, instrumentation integrity, and clinical outcomes (symptom and function improvement) based on investigator and patient-based outcome assessments.

The primary objective of this study is to document and analyze the use of NanoBone products in acute trauma cases (as a stand-alone bone graft, or in combination with local bone only, no other bone graft substitute or biologic product used) and determine both radiographic success and clinical outcomes. All product related adverse events will be documented, tabulated, and summarized.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects at least 18 years old at the time of injury
2. Acute fractures, resulting from blunt or penetrating trauma

   * In the extremities or pelvis
   * Requiring surgery
   * Treated emergently, delayed or staged up to 4 weeks from the date of injury
   * Where bone grafting is clinically indicated

Exclusion Criteria:

1. Certain fracture locations (these apply to non-unions as well)

   * Hand - metacarpals, phalanges
   * Forefoot - metatarsals, phalanges
   * Skull
   * Spine
2. Fractures requiring definitive fracture stabilization beyond the initial 4 weeks from the date of injury
3. Pathologic fractures secondary to malignancy
4. Subjects unable to follow recommended post-operative plan and complete follow ups
5. Subjects unable to complete patient reported outcome measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the study will be drawn from the individual surgeons' practice. Patients will be among those already surgically treated for trauma but have not completed their standard of care follow-up as determined by the surgeon's practice. In addition, the surgeon had determined that the use of a NanoBone product was clinically necessary for the patient. The choice of a NanoBone product was independent of this research project. Only patients who have had NanoBone implanted and consent to participate and meet the inclusion-exclusion criteria will be included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic evidence of fracture healing | 2 weeks, 6 weeks, 3 months, 6 months
  AP and lateral x-rays

SECONDARY OUTCOMES:
Pain relief | 2 weeks, 6 weeks, 3 months, 6 months
  Visual Analog Scale (VAS) pain score at fracture site. 0-10 scale, lower score means less pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell D Kuhl, DO, Principal Investigator — SSM Health
Locations (1):
- SSM Health St. Mary's Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No